CLINICAL TRIAL: NCT00249990
Title: Phase II Study of Aerosolized Liposomal 9-Nitro-20 (S)- Camptothecin (L9NC) in Patients With Metastatic or Recurrent Cancer of the Endometrium
Brief Title: Phase II Study of Aerosolized Liposomal 9-Nitro-20 (S)- Camptothecin (L9NC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Claire Verschraegen, MD; Principal Investigator, University of New Mexico
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1102C
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2008-10

CONDITIONS: Corpus Uteri; Endometrial Cancer
Keywords: Uterus; Recurrent disease; Treatment; 9-Nitrocamptothecin; Endometrium
MeSH Terms: conditions — Endometrial Neoplasms; Recurrence | interventions — rubitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: 9-NC in aerosol reservoir — Dose: 0.4 mg/ml of 9-NC in aerosol reservoir for 60 minutes (= daily dose of 0.52 mg/m2/day) per day X5 every week, X8 weeks, then observe for 2 weeks. One course = 10 weeks (45-47).

SUMMARY:
The purposes of this study are:

1.1 To determine the efficacy of liposomal 9-Nitro-20 (S)-Camptothecin (L9NC) administered by aerosolization to patients with metastatic endometrial cancer.

1.2 To determine toxicity profile of L9NC administered by aerosolization for 5 consecutive days per week X 8 weeks, every 10 weeks.

1.3 To perform a pharmacology study of L9NC in the plasma and the lungs after aerosolization. A specific protocol will be written for this part.

DETAILED DESCRIPTION:
RATIONALE: Camptothecin (CPT) is a plant alkaloid isolated from Camptotheca acuminata in 1966. As a topoisomerase I inhibitor, it has powerful anticancer properties and has been used clinically in the treatment of a variety of cancers. It possesses significant toxicity, especially involving the bone marrow and gastrointestinal tract that has limited its use. Derivatives of 20-(S)-camptothecin have been made to increase the aqueous solubility of these compounds and/or modify the A-ring to increase membrane association. The 9-nitrocamptothecin (9-NC) derivative to be used in this study is insoluble in water, but has demonstrated potent antitumor effects in mice and antitumor effect in humans. However, the therapeutic index is low. In order to increase the therapeutic index, a liposomal formulation has been developed, which can be administered as an aerosol. In humans, dose of 0.52 mg/m2/day 5 days per weeks for eight 8 weeks of a 10 week course were well tolerated in the Phase I study. Partial responses were noted in patients with endometrial cancers. The recommended starting dose of L9NC in the Phase II study is 0.52 mg/m2/day to be administered once a day by aerosol (mouth-only breathing) for five consecutive days per week x 8 weeks followed by a 2 week rest. Courses are 10 weeks. This dose corresponds to approximately 1/6 of the MTD of oral 9-NC administered to untreated cancer patients.

ELIGIBILITY:
Inclusion criteria:

* All patients, 18 years of age or older, with metastatic and/or recurrent endometrial cancer or with mixed mesenchymal malignant tumors whose epithelial component is recurring, who have failed standard chemotherapy or hormonal regimens for their disease or who refuse recommended standard chemotherapy are eligible.
* Patients must have a life expectancy of at least 12 weeks.
* Patients must have a Zubrod performance status of 0-2.
* Patients must sign an informed consent.
* Patients should have adequate bone marrow function defined by an absolute peripheral granulocyte count of >1,500 cells/mm3 and platelet count >100,000/mm3 and absence of a regular red blood cell transfusion requirement.
* Patients should have adequate hepatic function with a total bilirubin < 2 mg/dl and SGOT or SGPT < two times the upper limit of normal, and adequate renal function as defined by a serum creatinine < 1.5 x upper limit of normal.
* Patients must not have a known symptomatic respiratory disease other than cancer, and must have a pulmonary function test equal to >50% forced expiratory volume in 1 second (FEV1), >50% FEV1/forced vital capacity (FVC), >50% total lung capacity (TLC), and >50% diffusing capacity of the lung for carbon monoxide (DLCO) of predicted values.

Exclusion Criteria:

* Patients with symptomatic brain metastases are excluded from this study.
* Pregnant women or nursing mothers are not eligible for this trial. Patients of child bearing potential must use adequate contraception.
* Patients may receive no other concurrent chemotherapy or radiation therapy during this trial.
* Patients with severe medical problems such as uncontrolled diabetes mellitus or cardiovascular disease or active infections are not eligible for this trial.
* Any criteria that is borderline and may lead to ineligibility will be reviewed by the principal investigator (PI), who may override the eligibility criteria, after receiving sponsor agreement, if entry into the study is deemed to potentially benefit the patient.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2003-04; Primary Completion 2006-07 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Overall response rate (complete and partial responses).Activity will be calculated as the proportion of pts with responsive disease & the 95% confidence interval for response. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Claire Verschraegen, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States